CLINICAL TRIAL: NCT03637049
Title: A Phase 1, Drug-Drug Interaction Study to Evaluate the Effect of PBI-4050 on the Pharmacokinetics of Midazolam, a Sensitive Cytochrome P450 3A Substrate, in Healthy Adult Subjects
Brief Title: Effect of PBI-4050 on the Pharmacokinetics of Midazolam in Heathy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Liminal BioSciences Ltd. (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PBI-4050-CT-9-16; CA25590 (Other: Celerion)
Record Dates: First submitted 2018-08-08; First posted 2018-08-17 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Healthy
Keywords: PBI-4050; drug-drug interaction; CYP3A; midazolam; healthy subjects
MeSH Terms: interventions — setogepram; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PBI-4050 and midazolam (Experimental): Midazolam 2 mg solution once (Period 1), PBI-4050 1200 mg (3 x 400 mg tablets) once per day for 5 days and midazolam 2 mg solution once on last day (Period 2).
  Interventions: Drug: PBI-4050 and midazolam

INTERVENTIONS:
Drug: PBI-4050 and midazolam — A single oral dose of midazolam (1 mL of 2mg/mL syrup) will be given to all subjects in Period 1 and on Day 5 of Period 2. 1200 mg of PBI-4050 (3 X 400 mg tablets) will be administered for 5 days (Day 1 to Day 5) of Period 2 and a single dose of midazolam (1 mL of 2mg/mL) on Day 5.

SUMMARY:
This study is designed to evaluate the pharmacokinetics (PK) and safety of multiple doses of PBI-4050 combined with midazolam in healthy adult subjects.

DETAILED DESCRIPTION:
This is a Phase 1, single-center, open-label, 2-period, fixed sequence study to investigate the effect of multiple doses of PBI-4050 on the PK of midazolam, a cytochrome P450 (CYP) 3A substrate, in healthy adult men and healthy women of non-childbearing potential (WONCBP), and to determine the safety and tolerability of PBI-4050, when co-administered with midazolam.

On Day 1 of Period 1, subjects will receive a single oral dose of midazolam followed by PK sampling of midazolam and its metabolite 1-hydroxymidazolam (1-OH-midazolam). In Period 2, subjects will receive multiple daily doses of PBI-4050 for 5 consecutive days (Day 1 to Day 5) with a single oral dose of midazolam co-administered on Day 5. PK sampling for midazolam and 1-OH-midazolam will be collected for 24 hours following dosing on Day 5. PK sampling for PBI-4050 and its major metabolite will be collected at pre-dose on Days 3, 4, and 5.

There will be a washout period of at least 2 days between midazolam dose in Period 1 and the first PBI-4050 dose in Period 2.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females (WONCBP only).
2. Age 18-65 years.
3. Continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to the first dosing.
4. Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2 at screening.
5. Generally good health.
6. Males willing to use appropriate contraception.

Exclusion Criteria:

1. Significant medical history or physical findings.
2. History or presence of drug allergy or hypersensitivity to treatment ingredients.
3. Gastrointestinal surgery.
4. Pregnant or lactating.
5. Positive urine drug or alcohol screen.
6. Abnormal heart rate or blood pressure.
7. Prescribed systemic or topical medication taken recently, or supplements/remedies interfering with study procedures or safety.

   • Receiving drugs known as significant inducers of CYP2C9, CYP3A4, CYP2C8 and/or CYP1A2 enzymes and/or P-glycoprotein, including St. John's Wort, for 28 days prior to the first dosing and throughout the study.
8. Has been on a diet incompatible with the on-study diet.
9. Recent blood donation or significant blood loss.
10. Recent blood received.
11. Participation in another clinical study within 30 days prior to the first.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Change in area under the concentration-time curve (AUC0-t) for midazolam and 1-OH-midazolam in presence of PBI-4050 | PK sampling at pre-dose; and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours post-dose on Day 1 in Period 1 and on Day 5 in Period 2
  AUC0-t (AUC from time 0 to last observed non-zero concentration) of midazolam and 1-OH-midazolam assessed on Day 1 (Period 1) and Day 5 (Period 2)
Change in area under the concentration-time curve (AUC0-inf) for midazolam and 1-OH-midazolam in presence of PBI-4050 | PK sampling at pre-dose; and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours post-dose on Day 1 in Period 1 and on Day 5 in Period 2
  AUC0-inf (AUC from time 0 extrapolated to infinity) of midazolam and 1-OH-midazolam assessed on Day 1 (Period 1) and Day 5 (Period 2)
Change in maximum plasma concentration (Cmax) for midazolam and 1-OH-midazolam in presence of PBI-4050 | PK sampling at pre-dose; and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours post-dose on Day 1 in Period 1 and on Day 5 in Period 2
  Cmax of midazolam and 1-OH-midazolam assessed on Day 1(Period 1) and Day 5 (Period 2)
Change in concentration observed at the end of the dosing interval (Ctrough) for plasma PBI-4050 and its major metabolite | PK sampling for PBI-4050 and its metabolite done at pre-dose on Days 3, 4, and 5 of Peiod 2
  Ctrough is the concentration observed at the end of the dosing interval in Period 2.

SECONDARY OUTCOMES:
Adverse Events (AEs) and Serious Adverse Events (SAEs) | 10 days
  Number of subjects that experience Adverse Events (AEs).

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data for all primary and secondary outcome measures may be made available upon request.